CLINICAL TRIAL: NCT02234947
Title: Pancreas Volume in Preclinical Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Diabetes Action Research and Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600705 - N; 89-2013 (Other: Legacy study); DP3DK101120 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; pancreas volume
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Magnetic Resonance Spectroscopy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- New onset of Type 1 Diabetes: The subjects with new onset of Type 1 Diabetes will have pancreatic volume assessment by ultrasonography (US), Magnetic Resonance Imaging (MRI) and biochemical testing. These test will be compared to the testing from the other groups.
  Interventions: Procedure: MRI, US, and blood samples
- Antibody Positive Risk for Diabetes: The subjects with single or double antibody positive risk for Type 1 Diabetes will have pancreatic volume assessment by ultrasonography (US), Magnetic Resonance Imaging (MRI) and biochemical testing. These test will be compared to the testing from the other groups.
  Interventions: Procedure: MRI, US, and blood samples
- Antibody Negative Risk for Diabetes: The subjects with antibody negative risk for Type 1 Diabetes will have pancreatic volume assessment by ultrasonography (US), Magnetic Resonance Imaging (MRI) and biochemical testing. These test will be compared to the testing from the other groups.
  Interventions: Procedure: MRI, US, and blood samples
- Healthy Control: The subjects has no family history for Type 1 Diabetes. They will have pancreatic volume assessment by ultrasonography (US), Magnetic Resonance Imaging (MRI) and biochemical testing. These test will be compared to the testing from the other groups.
  Interventions: Procedure: MRI, US, and blood samples

INTERVENTIONS:
Procedure: MRI, US, and blood samples — All groups will have pancreatic volume assessment by ultrasonography (US), Magnetic Resonance Imaging (MRI) and blood samples. These test will be compared to the testing from the other groups.
  Other Names: Magnetic Resonance Imaging; Ultrasounography

SUMMARY:
Type 1 diabetes (T1D) is characterized by a progressive destruction of insulin producing beta cells, resulting in a lifelong dependence on exogenous insulin. While beta cells make up less than 1% of the pancreas, studies have demonstrated that T1D is associated with a marked reduction of pancreatic mass at diagnosis and as the disease progresses. As such, if pancreatic volume assessment, by ultrasonography (US) or MRI (Magnetic Resonance Imaging), could be utilized as a marker of beta cell function in high risk patients, non-invasive pancreatic imaging could become an important part of staging diabetes risk. As such, the primary goal of this study is to measure pancreatic volume and compare differences in volume between new onset T1D patients, antibody positive subjects at risk for diabetes, antibody negative individuals, and healthy controls.

DETAILED DESCRIPTION:
Participants will have blood tests and two imaging tests. The blood tests will tell us how well the pancreas is working. The imaging tests will measure the volume of the pancreas. There is one study visit associated with this study.

Blood will be drawn for 5 different blood tests. The participant cannot eat or drink for about 8 hours before the blood test (water is allowed). The blood will be sent to a lab. The amount of blood taken is equal to about 1 table spoon. Here are the blood tests that will be performed:

1. C-peptide - is used to measure the insulin being made by the cells in the pancreas.
2. Hemoglobin A1c (HbA1c) - is a measure of blood sugar control over the last 2 to 3 months.
3. Serum trypsin - is used to measure exocrine pancreatic function.
4. Glucose - is used to measure the amount of blood sugar in your body.
5. Autoantibodies (diabetes related) - are proteins that are made by the body's immune system. They are a sign that the cells in the pancreas that produce insulin could be damaged.

For the imaging procedures the participant cannot eat for at least 8 hours before the imaging procedure (water is okay). Your empty stomach will allow us to picture the pancreas better.

1. Magnetic resonance imaging (MRI) is a procedure that allows doctors to look inside the body by using a scanner that sends out a strong magnetic field and radio waves but involves no radiation exposure.
2. Ultrasound (US) is a device that consists of computer and a transducer that is used to scan the body. A transducer is a small hand-held device about the size of a bar of soap that is attached to the scanner by a cord. A lubricating gel is spread on the skin over the area being examined, and then the transducer is pressed firmly against the skin to obtain images.

These imaging tests will allow us to measure the volume of your pancreas. You will not get any sedation for these tests. If you cannot tolerate the MRI, then we will only do the US.

ELIGIBILITY:
Inclusion Criteria:

* T1D must be diagnosed less than one year
* Antibody status is know because of participation in TrialNet
* Healthy Control has no history or family history of T1D or other autoimmune disease

Exclusion Criteria:

* T1D diagnosis more than one year
* Antibody satus is not know
* Healthy Control has a family history of autoimmune disease
* unable to tolerate MRI and ultrasound

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The new onset will be people that have been diagnosed with T1D for less than one year. The anitbody negative or anitbody positive will be people that have been enrolled in the TrialNet study, Pathway to Prevention. The healthy control will be people from the general population with no history or family history of T1D.
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2013-11; Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
MRI of Pancreatic volume | Baseline
  Participants will undergo an MRI of their pancreas for volume assessment.
Ultrasound of Pancreatic volume | Baseline
  Participants will undergo a ultrasound of their pancreas for volume assessment.

SECONDARY OUTCOMES:
Blood Test will be done for pancreatic function and diabetes markers | Baseline
  Blood samples will be done for the following test: A1c, C-peptide, pancreatic autoantibodies, serum chymotrypsinogen.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Haller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Atkinson MA. The pathogenesis and natural history of type 1 diabetes. Cold Spring Harb Perspect Med. 2012 Nov 1;2(11):a007641. doi: 10.1101/cshperspect.a007641. PMID 23125199
- [Background] Campbell-Thompson M, Wasserfall C, Montgomery EL, Atkinson MA, Kaddis JS. Pancreas organ weight in individuals with disease-associated autoantibodies at risk for type 1 diabetes. JAMA. 2012 Dec 12;308(22):2337-9. doi: 10.1001/jama.2012.15008. No abstract available. PMID 23232891
- [Derived] Ross JJ, Wasserfall CH, Bacher R, Perry DJ, McGrail K, Posgai AL, Dong X, Muir A, Li X, Campbell-Thompson M, Brusko TM, Schatz DA, Haller MJ, Atkinson MA. Exocrine Pancreatic Enzymes Are a Serological Biomarker for Type 1 Diabetes Staging and Pancreas Size. Diabetes. 2021 Apr;70(4):944-954. doi: 10.2337/db20-0995. Epub 2021 Jan 13. PMID 33441381
- [Derived] Campbell-Thompson ML, Filipp SL, Grajo JR, Nambam B, Beegle R, Middlebrooks EH, Gurka MJ, Atkinson MA, Schatz DA, Haller MJ. Relative Pancreas Volume Is Reduced in First-Degree Relatives of Patients With Type 1 Diabetes. Diabetes Care. 2019 Feb;42(2):281-287. doi: 10.2337/dc18-1512. Epub 2018 Dec 14. PMID 30552130